CLINICAL TRIAL: NCT04075669
Title: Multiplex Strip PCR for Valid, Fast and Comprehensive Multi-pathogen Detection to Support the Diagnosis of Eye Infection Diseases (Endophthalmitis, Keratitis, Corneal Ulcers) From Corneal Scraping Samples
Brief Title: Multiplex Strip Polymerase Chain Reaction for Diagnosis of Eye Infection Diseases From Corneal Scraping Samples
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Made Susiyanti, Dr., dr., SpM(K), Research Coordinator, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Other Study IDs: 19-06-0699
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Endophthalmitis; Keratitis; Corneal Ulcer; Eye Infections
Keywords: Multiplex solid-phase strip PCR; Eye Infections; Endophthalmitis; Corneal Ulcer; Keratitis; Corneal Scraping Samples
MeSH Terms: conditions — Endophthalmitis; Keratitis; Corneal Ulcer; Eye Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Corneal scraping samples that will have its DNA extracted
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiplex Strip PCR — Corneal scraping from patients will have its DNA extracted and eluted in the buffer. The DNA than mixed with the primer strips tube and be analyzed in Real-Time PCR machine. According to the record information from the hospital, the pathogen that usually found from endophthalmitis, keratitis, corneal ulcer diseases in our hospital is Pseudomonas sp., Staphylococcus aureus, Staphylococcus epidermidis, Acinetobacter sp., Pseudomonas aeruginosa, Acanthamoeba sp., Aspergillus fumigatus, Aspergillus flavus, Fusarium sp., and Candida albicans. And based on the report from Zhao et al (2014) Herpes Simplex Virus may be detected from patients with keratitis. Therefore in this study, we are trying to detect all of the pathogens simultaneously using the real-time PCR assay from patients corneal scraping who experience eye infections as mention above.

SUMMARY:
The aim of this study is to see if multiplex strip PCR will detect the pathogen that causing eye infection from the corneal scraping samples with higher sensitivity and specificity than the current gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Registered as new patients since July 2019 in RSCM Kirana
* Age more than 18 years
* Have an eye infection (keratitis, endophthalmitis and corneal ulcer) which required corneal scrapping sampling for further diagnosis

Exclusion Criteria:

- Not willing to become the participants by not filling the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eye infections (Keratitis, endophthalmitis, and corneal ulcer) in RSCM Kirana Infection and Immunology Division that registered since July 2019
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Higher sensitivity and specificity by multiplex strip PCR than current gold standard | 4 months
  Ferrer and Alio (2011) report from 10 years of study shown that culture test as current gold standard will provide positive value by 59.3% for detecting keratitis pathogen. Based on this report, we see the potential increase of positive value by using multiplex PCR around 20 points (70%). Sensitivity will be calculated by true positive divided by all positive patients and specificity will be calculated by true negative divided by all negative patients. The results will be compared with the current gold standard with target increase 20 points or 70%.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. dr. Made Susiyanti, Sp.M(K), Principal Investigator — Infection and Immunology Department of Ophthalmology Faculty of Medicine Universitas Indonesia
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta Pusat, DKI Jakarta, Indonesia